CLINICAL TRIAL: NCT01958918
Title: A 12-month, Phase IV, Randomized, Open Label, Multicenter Study to Compare Efficacy of 0.5 mg Ranibizumab Pro re Nata (PRN) Versus 2 mg Aflibercept Bimonthly Intravitreal Injections on Retinal Thickness Stability Till Month 6 of Treatment and Explore Functional Outcomes up to Month 12 in Patients With Neovascular (Wet) Age-related Macular Degeneration (AMD)
Brief Title: Efficacy of Ranibizumab Prn Treatment Compared to Aflibercept Bimonthly Intravitreal Injections on Retinal Thickness Stability in Patients With Wet AMD
Acronym: SALT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002ADE23
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-12

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: wet age-related macular degeneration (AMD); ranibizumab; aflibercept; Best Corrected Visual Acuity (BCVA); Spectral Domain Optical Coherence Tomography (SD-OCT)
MeSH Terms: interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The reading center was masked for treatment assignment in order to ensure unbiased evaluation of the primary, secondary and exploratory objectives that were determined by SDOCT, autofluorescence imaging, and microperimetry and multifocal ERG (where available).
  When communicating with the reading center study centers had to be vigilant not to unblind the reading center to the treatment.
  Site staff performing the assessments of BCVA, contrast sensitivity (where possible), VFQ25 and IReST (reading speed) were also masked to the identity of the treatment.
  The central laboratory used for analysis of all specimens collected for biomarker assessment were blinded to the identity of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranibizumab (Experimental): 1 intravitreal injection monthly until maximum stable BCVA with retreatment based on BCVA loss and/or SD-OCT signs of wet AMD disease activity
  Interventions: Drug: Ranibizumab
- Aflibercept (Active Comparator): 1 intravitreal injection monthly for the first 3 months, followed by 1 intravitreal injection every 2 months
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Ranibizumab — 0.5 mg intravitreal injection
  Other Names: Lucentis®
  Arms: Ranibizumab
Drug: Aflibercept — 2 mg intravitreal injection
  Other Names: Eylea®
  Arms: Aflibercept

SUMMARY:
The purpose of this study was to compare the efficacy of 0.5 mg ranibizumab versus 2 mg aflibercept bimonthly intravitreal injections on retinal thickness stability.

DETAILED DESCRIPTION:
Patients attended 14 scheduled study visits during 12 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Visual impairment predominantly due to neovascular AMD Active
* Newly diagnosed, untreated, angiographically documented choroidal neovascularization (CNV) lesion

Key Exclusion Criteria:

* Stroke or myocardial infarction less than 3 Months prior to study entry
* Active injection or inflammation of either eye at the time of study entry
* Any type of systemic disease (or received treatment for it), including any medical condition (controlled or uncontrolled) that were to be expected to progress, recur, or change to an extent which could bias the assessment of the clinical status of the patient to a significant degree or put the patient at special risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2013-10-23 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2017-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (59):
- Austria (5):
  - Novartis Investigative Site, Feldkirch
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Laken
  - Novartis Investigative Site, Leuven
- Denmark (2):
  - Novartis Investigative Site, Glostrup Municipality
  - Novartis Investigative Site, Roskilde
- France (3):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Paris
- Germany (31):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Bad Rothenfelde
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Glauchau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Siegburg
  - Novartis Investigative Site, Sulzbach
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wolfsburg
  - Novartis Investigative Site, Würzburg
- Netherlands (3):
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Nijmegen
- Norway (2):
  - Novartis Investigative Site, Arendal
  - Novartis Investigative Site, Oslo
- Portugal (6):
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Vila Franca de Xira
  - Novartis Investigative Site, Vila Nova de Gaia
- Sweden (2):
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Västerås
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Fribourg
  - Novartis Investigative Site, Geneva

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 6 sites in Austria, 2 sites in Belgium, 2 sites in Denmark and 5 sites from France.
Pre-assignment Details: This reporting group included all patients randomized to one of the treatment arms (Randomized Set)
  The Full Analysis Set (FAS) consisted of all patients who received at least one application of study treatment and had at least one post-baseline assessment for SD-OCT.
Groups:
- Ranibizumab: 0.5 mg intravitreal injections of ranibizumab monthly until maximum stable BCVA with retreatment based on BCVA loss and/or SD-OCT signs of wet AMD disease activity.
- Aflibercept: 2 mg intravitreal injections of aflibercept monthly for the first 3 months, followed by 2 mg intravitreal injections once every 2 months (current EU SmPC label)
Period: Overall Study
Arm/Group | Ranibizumab | Aflibercept
Started (patients randomized) | 356 | 356
Full Analysis Set | 353 | 354
Completed (completed overall) | 313 | 314
Not Completed | 43 | 42
Not completed — Death | 1 | 3
Not completed — Lost to Follow-up | 4 | 7
Not completed — Withdrawal by Subject | 13 | 8
Not completed — Lack of Efficacy | 13 | 10
Not completed — Adverse Event | 12 | 12
Not completed — administrative problems | 0 | 2

BASELINE CHARACTERISTICS:
Population: FAS
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab | Aflibercept | Total
Number analyzed (Participants) | 353 | 354 | 707
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.3 (7.53) | 78.0 (7.21) | 77.7 (7.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 218 | 428
  Male | 143 | 136 | 279
Race/Ethnicity, Customized [Number; unit: Participants] — Population: FAS
  Participants
    Caucasian | 350 | 352 | 702
    Asian | 1 | 0 | 1
    Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean of the Absolute Values of CSRT Difference Month 3 to Month 6
Description: The thickness of the retina was measured by Spectral Domain Optical Coherence Topography (SD-OCT). The mean of the absolute values of the CSRT difference between Month 3 and 4, Month 4 and 5, and Month 5 and 6 was calculated (ie, CSRT fluctuation). A lower average CSRT fluctuation demonstrates greater retinal stability. One eye (study eye) contributed to the analysis.
Time Frame: Month 3, Month 4, Month 5, Month 6
Population: FAS. Number analyzed is the number of patients with a measurement
Measure: Mean (Standard Error); unit: micrometers
Arm/Group | Ranibizumab | Aflibercept
Number analyzed (Participants) | 345 | 340
micrometers | 25.16 (2.584) | 29.28 (2.620)
Statistical Analysis 1: Comparison: Ranibizumab vs Aflibercept; Test type: Superiority; p = 0.1850, ANOVA

2. Secondary Outcome: Total Best Corrected Visual Acuity (BCVA) Score Measured in ETDRS Letters at Month 12
Description: Visual acuity was assessed in a sitting position with refraction using ETDRS-like visual acuity testing charts at an initial testing distance of 4 meters. A higher score indicates better visual acuity. ETDRS scale ranges from 0-100 letters. A score of 65 to 70 letters represents a low to moderate visual acuity
Time Frame: Month 12
Population: FAS with measurement at visit Month 12. No statistical analysis was performed.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab | Aflibercept
Number analyzed (Participants) | 313 | 312
letters | 66.4 (18.10) | 68 (17.62)

3. Secondary Outcome: IREST at Month 12
Description: Number of incorrectly read words (IREST) was assessed using International Reading Speed Texts (IResT) and measured in words per minute.
Time Frame: Month 12
Population: FAS with measurement at Month 12. No statistical analysis was performed.
Measure: Mean (Standard Deviation); unit: incorrect words per minute
Arm/Group | Ranibizumab | Aflibercept
Number analyzed (Participants) | 253 | 251
incorrect words per minute | 5.7 (21.19) | 6.1 (21.86)

4. Secondary Outcome: National Eye Institute Visual Functioning Questionnaire Composite Score (VFQ-25) at Month 12
Description: Vision-related quality of life was assessed by the patient using the National Eye Institute Visual Function Questionnaire. The scores of 12 subscales (general health, general vision, ocular pain, near activities, distance activities, social function, mental health, role difficulties, dependency, driving, color vision, and peripheral vision) were added together for a total (composite) score, which ranged from 0 to 100. A higher score indicates poorer function.
Time Frame: Month 12
Population: FAS with measurement at Month 12. No statistical analysis was performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab | Aflibercept
Number analyzed (Participants) | 305 | 297
units on a scale | 80.0 (14.43) | 79.1 (14.95)

5. Secondary Outcome: Correlations Between CSRT Fluctuation (Month 3 to 6) and Functional Outcomes at Month 12 (Full Analysis Set)
Description: Correlation coefficient calculated based on Pearson's correlation between each corresponding parameter and CSRT stability.
Time Frame: Month 3 to Month 6, Month 12
Population: Full Analysis Set with measure. No statistical analysis was performed.
Measure: Number; unit: correlation coefficient
Arm/Group | Ranibizumab | Aflibercept
Number analyzed (Participants) | 353 | 354
correlation coefficient
  Total BCVA Score: number analyzed (Participants) | 313 | 310
  Total BCVA Score | -0.2194 | 0.0155
  IREST reading speed (words/minute): number analyzed (Participants) | 252 | 249
  IREST reading speed (words/minute) | 0.0889 | 0.0450
  VFQ-25 composite score: number analyzed (Participants) | 306 | 295
  VFQ-25 composite score | 0.1064 | 0.0847

ADVERSE EVENTS:
Time Frame: 1 year
Description: AE additional description
Groups:
- Ranibizumab 0.5 mg: Ranibizumab 0.5 mg
- Aflibercept 2 mg: Aflibercept 2 mg
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2 mg
All-Cause Mortality (participants affected / at risk) | 1/356 | 3/356
Serious Adverse Events (participants affected / at risk) | 67/356 | 74/356
Other Adverse Events (participants affected / at risk) | 156/356 | 156/356
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=356) | Aflibercept 2 mg (N=356)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 5
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 3 | 4
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 1
Systolic dysfunction (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Amaurosis fugax (Eye disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Detachment of macular retinal pigment epithelium (Eye disorders) | 0 | 1
Ectropion (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Iridocyclitis (Eye disorders) | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 2
Retinal pigment epithelial tear (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Vitreous adhesions (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 3
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Medical device site joint pain (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Abscess oral (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Endophthalmitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Lip infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 3
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Body temperature decreased (Investigations) | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Fluid retention (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Akinesia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Brain stem stroke (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 3 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 3 | 3
Cervical myelopathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Formication (Nervous system disorders) | 1 | 0
Glossopharyngeal neuralgia (Nervous system disorders) | 1 | 0
Hyperkinesia (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 2
Vascular dementia (Nervous system disorders) | 0 | 1
Device breakage (Product Issues) | 0 | 1
Emotional distress (Psychiatric disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Urethral dilatation (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 2
Hypertensive crisis (Vascular disorders) | 4 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=356) | Aflibercept 2 mg (N=356)
Conjunctival haemorrhage (Eye disorders) | 41 | 28
Dry eye (Eye disorders) | 18 | 11
Eye pain (Eye disorders) | 24 | 23
Ocular hyperaemia (Eye disorders) | 20 | 9
Visual acuity reduced (Eye disorders) | 19 | 25
Influenza (Infections and infestations) | 22 | 12
Viral upper respiratory tract infection (Infections and infestations) | 43 | 62
Intraocular pressure increased (Investigations) | 29 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 21
Hypertension (Vascular disorders) | 16 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and condition of Novartis'agreements with its investigator may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.